CLINICAL TRIAL: NCT06949540
Title: A Clinical Trial to Evaluate the Effects of a Herbal Tincture on Energy Levels, Weight Management, and Markers of Metabolic Health
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Apothekary (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20716
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Stress; Fatigue
Keywords: Weight Management; Energy Levels
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blue Burn Tincture Group (Experimental): Participants will receive 4 mL of the Blue Burn Tincture daily for 12 weeks. The dose is split into 2 mL in the morning and 2 mL at lunchtime (before 2 PM), mixed with water or another liquid.
  Interventions: Dietary Supplement: Blue Burn Tincture

INTERVENTIONS:
Dietary Supplement: Blue Burn Tincture — Participants will complete self-assessments and provide weight and blood measurements during the study.

SUMMARY:
This study will evaluate the effects of the Blue Burn Tincture on energy levels, weight management, and markers of metabolic health. It is a single-arm, hybrid trial involving 40 participants over a 12-week period. Participants will use the product daily, complete scheduled questionnaires, attend blood tests at Labcorp (Baseline and Week 12), and provide body mass measurements. Primary outcomes include changes in cortisol levels, energy levels, and body mass.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female.
* Be aged 30 or over.
* Anyone who owns a body weight scale.
* Anyone currently experiencing issues regarding all of the following:

  1. Self-reported feelings of stress.
  2. Self-reported issues with maintaining their current body weight or losing weight.
* Exercises at least once per week.
* If taking prescription medications, are willing to discuss this study with their physician before starting the study.
* Willing to maintain the study protocol for the study duration.
* Willing to refrain from taking any products, new medication, or supplements that target cortisol levels, stress, energy levels, or weight management during the study duration.
* If taking oral over-the-counter supplements or herbal remedies targeted at improving cortisol levels, stress, energy levels, or weight management, has been consistently taking these for at least 3 months prior to starting the study and is willing to maintain this routine for the study duration.
* Willing to maintain their current diet, sleep schedule, and activity level for the study duration.
* Anyone who is generally healthy - does not live with any uncontrolled chronic disease.
* Resides in the United States.
* Not currently partaking in another research study and will not be partaking in any other research study for the next 12 weeks and at any point during this study's duration.

Exclusion Criteria:

* Anyone with pre-existing chronic conditions that would prevent participants from adhering to the protocol, including oncological and psychiatric disorders.
* Anyone who is planning to undergo any surgeries or invasive treatments for the study duration.
* Anyone diagnosed with a condition related to the thyroid.
* Anyone diagnosed with Type I or Type II diabetes.
* Anyone who has had any major illness in the last three months.
* Anyone who drinks heavily (i.e., eight or more alcoholic drinks per week for women or 15 or more alcoholic drinks per week for men).
* Anyone with an allergy to nightshade vegetables.
* Anyone with known severe allergic reactions to any of the study product ingredients.
* Any women who are pregnant, breastfeeding, or trying to conceive (or who will be at any point during the study period).
* Anyone with a history of substance abuse.
* Anyone who is currently a smoker or has been a smoker in the past 3 months.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-07 (Actual); Primary Completion 2025-05-07 (Estimated); Study Completion 2025-05-07 (Estimated)

PRIMARY OUTCOMES:
Change in cortisol levels | Baseline and Week 12
  Measured via morning blood draws at Baseline and Week 12 to assess the physiological impact of the tincture on stress hormone regulation.
Change in body mass | Baseline and Week 12
  Self-reported daily body mass measurements for 3 days at Baseline and Week 12; mean values will be calculated to determine any weight changes.
Change in self-reported energy levels | Baseline, Week 2, Week 4, Week 8, and Week 12
  Participants will complete validated questionnaires evaluating energy at multiple time points to assess perceived improvements in fatigue and vitality.

SECONDARY OUTCOMES:
Change in perceived workout performance and health metrics | Baseline, Week 2, Week 4, Week 8, and Week 12
  Questionnaires will assess participant perceptions of workout performance, stamina, exercise recovery, weight management, fitness, and overall health.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: Undecided